CLINICAL TRIAL: NCT06959966
Title: Effects of Oligo-fucoidan on Leiomyoma Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Hi-Q Marine Biotech International, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N201812056
Record Dates: First submitted 2025-03-14; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-03

CONDITIONS: Uterine Leiomyoma
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Starch capsule, 4 grams per day (two capsules), taken orally for six months. Capsules match the treatment group in odor and weight.
  Interventions: Combination Product: Placebo
- Treatment (Experimental): Oligo-Fucoidan capsule, 4 grams per day (two capsules), taken orally for six months.
  Interventions: Combination Product: Oligo Fucoidan

INTERVENTIONS:
Combination Product: Placebo — Starch capsule, 4 grams, two capsules per day for six months.
  Arms: Placebo
Combination Product: Oligo Fucoidan — Oligo fucoidan capsule, 4 grams, two capsules per day for six months.
  Arms: Treatment

SUMMARY:
Uterine leiomyoma is the most common benign tumor in women, with an incidence rate of approximately 20% among women of reproductive age. Patients may experience severe abdominal pain, abnormal bleeding, and infertility. Pathological examination of uterine specimens reveals that up to three-quarters of cases involve uterine leiomyoma, indicating that this condition is often accompanied by other uterine pathologies. Therefore, medical intervention remains necessary for affected patients. Currently, the most common treatment options include medication and surgical removal. However, the severe side effects of drug therapy and the high recurrence rate following surgical excision significantly impact patients' quality of life, underscoring the need for continued research into better treatment strategies. Fucoidan, a commercially available dietary supplement, has been shown in numerous studies to provide adjunctive therapeutic benefits for cancer patients. However, no clinical trials have been conducted to evaluate the effects of fucoidan on patients with uterine leiomyoma. Therefore, this clinical study aims to investigate the effects of fucoidan on patients with uterine leiomyoma.

ELIGIBILITY:
Inclusion Criteria:

* Women with uterine fibroids aged 20-55 years.
* Confirmation of uterine fibroids by ultrasound (more than 3 cm, less than 10 cm).
* There are no plans for pregnancy in the past six months.
* There were no plans for uterine fibroid surgery for nearly six months.
* Agree to abide by the research regulations.

Exclusion Criteria:

* A patient with heart disease, liver disease, kidney disease or any mental illness.
* Patients who are unable to communicate or criticize.
* Pregnant women.
* Patients taking regular medications, including serotonin, antidepressants or other antipsychotics.
* Non-native speakers.

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Leiomyoma patients
Enrollment: 18 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Leiomyoma Size | 6 months
  the size of leiomyoma tissue (mm)
Change in Number of Leiomyomas | 6 months
  the number of leiomyoma tissue

SECONDARY OUTCOMES:
Change in Triglyceride Level | 6 months
  TG (triglycerides): mg/dL
Change in Total Cholesterol Level | 6 months
  T-CHO (total cholesterol): mg/dL
Change in HDL Cholesterol Level | 6 months
  HDL-C (high-density lipoprotein cholesterol): mg/dL
Change in LDL Cholesterol Level | 6 months
  LDL-C (low-density lipoprotein cholesterol): mg/dL
Change in White Blood Cell Count | 6 months
  WBC (white blood cells), Unit: 10³/μL
Change in Red Blood Cell Count | 6 months
  RBC (red blood cells), Unit: 10⁶/μL
Change in Hemoglobin Level | 6 months
  HGB (hemoglobin) Unit: g/dL
Change in Hematocrit | 6 months
  HCT (hematocrit) Unit: %
Change in Blood Glucose | 6 months
  Measurement: AC (blood glucose) Unit: mg/dL
Change in High-Sensitivity C-Reactive Protein | 6 months
  High-Sensitivity C-Reactive Protein (HS-CRP) Unit: mg/dL
Change in Aspartate Aminotransferase | 6 months
  Aspartate Aminotransferase(AST) Unit: U/L
Change in Alanine Aminotransferase | 6 months
  Alanine Aminotransferase (ALT) Unit: U/L
Change in Blood Urea Nitrogen | 6 months
  Blood Urea Nitrogen (BUN) Unit: mg/dL
Change in Follicle-Stimulating Hormone | 6 months
  Follicle-Stimulating Hormone(FSH) Unit: mIU/mL
Change in Albumin | 6 months
  Albumin (ALB) Unit: g/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical Univeersity, Taipei, Xinyi, Taiwan

IPD SHARING:
Plan to Share IPD: No